CLINICAL TRIAL: NCT01370811
Title: A Phase II, Double-blind, Randomized, Placebo-controlled 4-way Crossover Study to Evaluate the Relative Efficacy and Safety of OC Oral Solution (Oxybutynin and Clonidine) for Sialorrhoea in Patients With Parkinson's Disease
Brief Title: A Relative Efficacy and Safety Study of OC Oral Solution for Sialorrhoea in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Orient Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OP-014-201
Record Dates: First submitted 2011-06-08; First posted 2011-06-10 (Estimated); Results first posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Sialorrhoea
Keywords: oxybutynin; clonidine; OC Oral Solution; sialorrhoea; Parkinson's disease
MeSH Terms: conditions — Sialorrhea; Parkinson Disease | interventions — oxybutynin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- oxybutynin and clonidine oral solution treatment D (Placebo Comparator): Placebo
  Interventions: Drug: oxybutynin and clonidine oral solution treatment D
- oxybutynin and clonidine oral solution treatment C (Experimental): High dose oxybutynin and clonidine
  Interventions: Drug: oxybutynin and clonidine oral solution treatment C
- oxybutynin and clonidine oral solution treatment A (Experimental): Low dose oxybutynin and clonidine
  Interventions: Drug: oxybutynin and clonidine oral solution treatment A
- oxybutynin and clonidine oral solution treatment B (Experimental): Intermediate dose oxybutynin and clonidine
  Interventions: Drug: oxybutynin and clonidine oral solution treatment B

INTERVENTIONS:
Drug: oxybutynin and clonidine oral solution treatment A
  Other Names: OP-014
  Arms: oxybutynin and clonidine oral solution treatment A
Drug: oxybutynin and clonidine oral solution treatment B
  Other Names: OP-014
  Arms: oxybutynin and clonidine oral solution treatment B
Drug: oxybutynin and clonidine oral solution treatment C
  Other Names: OP-014
  Arms: oxybutynin and clonidine oral solution treatment C
Drug: oxybutynin and clonidine oral solution treatment D — Placebo
  Other Names: Placebo
  Arms: oxybutynin and clonidine oral solution treatment D

SUMMARY:
The purpose of this study is to determine whether OC (oxybutynin and clonidine) oral solution is effective in reducing saliva secretion in patients suffering from Parkinson's Disease with excessive salivation.

DETAILED DESCRIPTION:
Sialorrhea is excessive flow of saliva associated with its unintentional loss from the mouth, commonly known as drooling. Sialorrhea may result from any combination of hypersecretion, problems swallowing or sensorimotor problems containing saliva in the mouth. It is commonly found in people with neurological dysfunction such as Parkinson's Disease, leading to social isolation and embarrassment. In general, treatment options are limited because of the underlying chronic disease. The objective of the proposed low-dose, new combination drug, OC Oral solution is to develop a new treatment option that can be used to titrate saliva secretion rates to a level that is low enough to prevent unintentional loss (i.e. drooling) but not so low as to cause an uncomfortably dry mouth.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's Disease for at least 2 years
* Patients with a score of ≥2 on the salivation section of UPDRS, item 6
* Patients Hoehn and Yahr stage must be ≤4
* under stable anti-Parkinson therapy throughout the study
* Able and willing to comply with the study procedures
* Able to provide and provision of a written informed consent

Exclusion Criteria:

* Female who is pregnant/lactating or planning to be pregnant
* Must not have a form of drug-induced or atypical parkinsonism or parkinsonism with swallow problems due to other etiology
* Have current uncontrolled hypertension, symptomatic postural hypotension, active Raynaud's disease or other peripheral vascular occlusive disease
* Have a history or presence of hyperthyroidism, congestive heart failure, coronary heart disease, cardiac arrhythmias, tachycardia or severe bradycardia resulting from either sick sinus syndrome or AV block of 2nd or 3rd degree
* Have a history of narrow angle glaucoma or shallow anterior chamber
* Have a history or presence of gastrointestinal obstruction, including paralytic ileus and intestinal atony or gastrointestinal motility disorders, toxic megacolon or severe ulcerative colitis
* Have a history or presence of bladder outflow obstruction or urinary retention
* Patients with hepatic or renal impairment
* Male with QTc > 430 ms or female with QTc > 450 ms ECG results at screening
* Concomitant use of α2-agonist, anticholinergic medication or other medications that affect ACh levels
* Have a history of alcohol or substance abuse
* Any condition, including the presence of laboratory abnormalities, which places the patient at unacceptable risk to participate in the study or confounds the ability to interpret data from the study
* Have a history of hypersensitivity to the investigational medicinal product or any of the excipients or to medicinal products with similar chemical structures
* Have received treatment with any other investigational medicinal product in the last 6 weeks before administration of the first dose in this clinical study
* Have received treatment with any medicinal product known to have a well-defined potential for toxicity to a major organ in the previous 3 months
* Have a positive result of the human immunodeficiency virus (HIV) 1 and 2 test
* Have problems to understand the protocol requirements, instructions and study related restrictions, the nature, scope and possible consequences of the clinical study
* Are unlikely to comply with the protocol requirements, instructions and study related restrictions
* Patient is the Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the clinical study
* Vulnerable subjects
* Have any concurrent disease or condition that, in the opinion of the Investigator, would make the patient unsuitable for participation in the clinical study
* Donation of 500 ml or more of blood within the last 8 weeks before start of the study and for at least 4 weeks after study completion
* Have previously been enrolled in this clinical study
* Vulnerable subjects

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron L Ellenbogen, DO, MPH, Principal Investigator — QUEST Research Institute; Chi-Tai Chang, PhD, Study Director — Orient Pharma Co., Ltd.
Locations (1):
- QUEST Research Institute, Bingham Farms, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This single center Phase II study was initated on 02 Aug 2011. First patient was screened on 25 Aug 2011. All the study patients were recruited from medical clinic and the patient recruitment ended on 23 Aug 2012.The last study patient completed study on 19 Sep 2012.
Pre-assignment Details: After informed consent process, investigators screened 35 patients and successfully randomized 24 patients to receive study treatments. The other 11 patients were screening failure since they failed to meet study required inclusion and/or exclusion criteria.
Groups:
- Sequence 1: Treatment A→Treatment B→Treatment D→Treatment C: Treatment A:Oxybutynin 2.0 mg and clonidine 37.5 μg Treatment B: Oxybutynin 5.0 mg and clonidine 50.0 μg Treatment C: Oxybutynin 7.5 mg and clonidine 75.0 μg Treatment D:Placebo
- Sequence 2: Treatment B→Treatment C→Treatment A→Treatment D: Treatment B: Oxybutynin 5.0 mg and clonidine 50.0 μg Treatment C: Oxybutynin 7.5 mg and clonidine 75.0 μg Treatment A:Oxybutynin 2.0 mg and clonidine 37.5 μg Treatment D:Placebo
- Sequence 3: Treatment C→Treatment D→Treatment B→Treatment A: Treatment C: Oxybutynin 7.5 mg and clonidine 75.0 μg Treatment D:Placebo Treatment B: Oxybutynin 5.0 mg and clonidine 50.0 μg Treatment A:Oxybutynin 2.0 mg and clonidine 37.5 μg
- Sequence 4: Treatment D→Treatment A→Treatment C→Treatment B: Treatment D:Placebo Treatment A:Oxybutynin 2.0 mg and clonidine 37.5 μg Treatment C: Oxybutynin 7.5 mg and clonidine 75.0 μg Treatment B: Oxybutynin 5.0 mg and clonidine 50.0 μg
Period: First Intervention
Arm/Group | Sequence 1: Treatment A→Treatment B→Treatment D→Treatment C | Sequence 2: Treatment B→Treatment C→Treatment A→Treatment D | Sequence 3: Treatment C→Treatment D→Treatment B→Treatment A | Sequence 4: Treatment D→Treatment A→Treatment C→Treatment B
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period of >=5 Days
Arm/Group | Sequence 1: Treatment A→Treatment B→Treatment D→Treatment C | Sequence 2: Treatment B→Treatment C→Treatment A→Treatment D | Sequence 3: Treatment C→Treatment D→Treatment B→Treatment A | Sequence 4: Treatment D→Treatment A→Treatment C→Treatment B
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Sequence 1: Treatment A→Treatment B→Treatment D→Treatment C | Sequence 2: Treatment B→Treatment C→Treatment A→Treatment D | Sequence 3: Treatment C→Treatment D→Treatment B→Treatment A | Sequence 4: Treatment D→Treatment A→Treatment C→Treatment B
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period of >=5 Days
Arm/Group | Sequence 1: Treatment A→Treatment B→Treatment D→Treatment C | Sequence 2: Treatment B→Treatment C→Treatment A→Treatment D | Sequence 3: Treatment C→Treatment D→Treatment B→Treatment A | Sequence 4: Treatment D→Treatment A→Treatment C→Treatment B
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Third Intervention
Arm/Group | Sequence 1: Treatment A→Treatment B→Treatment D→Treatment C | Sequence 2: Treatment B→Treatment C→Treatment A→Treatment D | Sequence 3: Treatment C→Treatment D→Treatment B→Treatment A | Sequence 4: Treatment D→Treatment A→Treatment C→Treatment B
Started | 6 | 6 | 6 | 6
Completed | 6 | 5 | 6 | 6
Not Completed | 0 | 1 | 0 | 0
Period: Washout Period of >=5 Days
Arm/Group | Sequence 1: Treatment A→Treatment B→Treatment D→Treatment C | Sequence 2: Treatment B→Treatment C→Treatment A→Treatment D | Sequence 3: Treatment C→Treatment D→Treatment B→Treatment A | Sequence 4: Treatment D→Treatment A→Treatment C→Treatment B
Started | 6 | 5 | 6 | 6
Completed | 6 | 5 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Fourth Intervention
Arm/Group | Sequence 1: Treatment A→Treatment B→Treatment D→Treatment C | Sequence 2: Treatment B→Treatment C→Treatment A→Treatment D | Sequence 3: Treatment C→Treatment D→Treatment B→Treatment A | Sequence 4: Treatment D→Treatment A→Treatment C→Treatment B
Started | 6 | 5 | 6 | 6
Completed | 6 | 5 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequence 1: Treatment A→Treatment B→Treatment D→Treatment C
- Sequence 2: Treatment B→Treatment C→Treatment A→Treatment D
- Sequence 3: Treatment C→Treatment D→Treatment B→Treatment A
- Sequence 4: Treatment D→Treatment A→Treatment C→Treatment B
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 3 | 4 | 13
  >=65 years | 4 | 2 | 3 | 2 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (6.46) | 64 (6.5) | 62 (7.45) | 62.8 (7.0) | 63 (7.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 1 | 7
  Male | 4 | 4 | 4 | 5 | 17
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Saliva Secreted Rate
Description: Change from baseline, negative mean reduce secret rate from baseline, positive mean not reduce secretion.
Time Frame: 8 hours post-dose
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Groups:
- OC Oral Solution Treatment B: Intermediate dose oxybutynin and clonidine
  OC oral solution treatment B :
- OC Oral Solution Treatment C: High dose oxybutynin and clonidine
  OC oral solution treatment C :
- OC Oral Solution Treatment D: Placebo
  OC oral solution treatment D : Placebo
- OC Oral Solution Treatment A: Low dose Oxybutynin and clonidine.
Arm/Group | OC Oral Solution Treatment B | OC Oral Solution Treatment C | OC Oral Solution Treatment D | OC Oral Solution Treatment A
Number analyzed (Participants) | 24 | 24 | 23 | 24
percentage of change from baseline | -6.508 (0.165) | -34.512 (0.147) | 83.695 (0.281) | 7.414 (0.175)

2. Secondary Outcome: Numeric Rating Scale (NRS) Measurements of Subjective Judgment of Excessive Saliva Production
Description: Evaluation of change from baseline the subjective assessment of saliva production after administration of a single dose of different combinations of oxybutynin and clonidine (OC Oral solution) in patients suffering from Parkinson's disease with excessive salivation. Compare with baseline the number of rate scale was more production with baseline or reduce from baseline.
  The min and max of the score is 0 and 10, the total range is 0~10, and higher value is represented more worse outcome.
Time Frame: 8 hours post-dose
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- OC Oral Solution Treatment A: Low dose oxybutynin and clonidine
  OC oral solution treatment A :
Arm/Group | OC Oral Solution Treatment A | OC Oral Solution Treatment B | OC Oral Solution Treatment C | OC Oral Solution Treatment D
Number analyzed (Participants) | 24 | 24 | 24 | 23
score on a scale | -0.8 (1.74) | -1.2 (1.71) | -1.6 (1.74) | -1.1 (1.83)

3. Secondary Outcome: Evaluation of the Safety and Tolerability of Different Combinations of Oxybutynin and Clonidine (OC Oral Solution) in Patients Suffering From Parkinson's Disease With Excessive Salivation
Description: Evaluation of the safety and tolerability of different combinations of oxybutynin and clonidine (OC Oral solution) in patients suffering from Parkinson's disease with excessive salivation. Calculate the treatment Emergent Adverse Events number during the study treatment period and follow up period up to at least 23 days excluding the screening period.
Time Frame: during the study treatment period and follow up period at least 23 days excluding the screening period.
Measure: Number; unit: Treatment Emergent Adverse Events
Groups:
- OC Oral Solution Treatment D: placebo oxybutynin and placebo clonidine
Arm/Group | OC Oral Solution Treatment A | OC Oral Solution Treatment B | OC Oral Solution Treatment C | OC Oral Solution Treatment D
Number analyzed (Participants) | 24 | 24 | 24 | 23
Treatment Emergent Adverse Events | 6 | 6 | 5 | 4

ADVERSE EVENTS:
Time Frame: 23 days for experimental period and follow up period.
Arm/Group | OC Oral Solution Treatment A | OC Oral Solution Treatment B | OC Oral Solution Treatment C | OC Oral Solution Treatment D
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 6/24 | 6/24 | 5/24 | 4/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OC Oral Solution Treatment A (N=24) | OC Oral Solution Treatment B (N=24) | OC Oral Solution Treatment C (N=24) | OC Oral Solution Treatment D (N=23)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Heart rate irregular (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to adverse event, one female patient (randomized number R24) did not complete her 4th study treatment (Treatment D/Placebo) in this 4-way cross over study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less